CLINICAL TRIAL: NCT04161352
Title: A Multicenter, Prospective Real World Study on Recombinant Human Endostatin (Endostar) Combined With Concurrent Radiochemotherapy for Treatment of Unresectable Stage III Non-small-cell Lung Cancer
Brief Title: Endostar Combined With Concurrent Radiochemotherapy for Treatment of Unresectable Stage III NSCLC
Acronym: R-helper
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Endo-CCRT-001
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Unresectable Stage III NSCLC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The chemoradiotherapy (CCRT) is still a standard treatment for the unresectabl stage III NSCLC.However, prognosis following this treatment is generally poor, with 5-year survival of 15-20%. The result of published HELPER study had showed that Endostar, a kind of angiogenesis agent, in combination with CCRT could improve the efficacy and safety. In order to verify the rusults, the investigators design the current study.

DETAILED DESCRIPTION:
The current study is a observation study in the real world setting. The 500 patients in compliance with Enrollment Criteria will be as the objects of observation. The procedure of study include the period of screening, treating and follow-up. The duration of study is about two and half year. The data entrying will be done by CRC, using the EDC system. CRA will audit the quality of data regularly.

ELIGIBILITY:
Inclusion Criteria:

* untreated pathologically confirmed inoperable stage III NSCLC according to the 8th edition of the American Joint Committee on Cancer staging system;
* at least one measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST)1.1;
* 18-75 years of age;
* Eastern Cooperative Oncology Group performance status score (ECOG PS) of 0 to 1;
* 10) FEV1>1.0 L;
* suitable function of bone marrow, liver, kidney and coagulation

Exclusion Criteria:

history of other malignant diseases, uncontrolled hypertension, any contraindications to chemoradiotherapy, pregnancy, breastfeeding or preexisting bleeding diatheses.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients with untreated pathologically confirmed inoperable stage III NSCLC, suitable for the treatment of CCRT
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-11-25 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 15 months
  progress free survival

SECONDARY OUTCOMES:
OS | 3 years
  Overall survival
LRFS | 2 years
  Locoregional relapse-free survival
DMFS | 2 years
  Distant metastasis-free survival
AEs | 3 years
  adverse events

IPD SHARING:
Plan to Share IPD: No
Only principlal investigator has the right to use all the data collected. The individual participant will not be allowed to share the data among them.